CLINICAL TRIAL: NCT05146531
Title: Comparison of McCoy Laryngoscope and C-MAC D-blade Video Laryngoscope in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun Young Park (Other)
Responsible Party: Sponsor-Investigator, Eun Young Park, Associate professor, Hallym University Medical Center
Organization: Hallym University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-10-010
Record Dates: First submitted 2021-11-18; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: obesity; intubation; laryngoscopes
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McCoy group (Active Comparator): Patients were intubated with McCoy laryngoscope.
  Interventions: Device: McCoy laryngoscope
- C-MAC group (Experimental): Patients were intubated with C-MAC D-blade video laryngoscope.
  Interventions: Device: C-MAC D-blade video laryngoscope

INTERVENTIONS:
Device: McCoy laryngoscope — Patients scheduled for general anesthesia were intubated with McCoy laryngoscope.
  Arms: McCoy group
Device: C-MAC D-blade video laryngoscope — Patients scheduled for general anesthesia were intubated with C-MAC D-blade video laryngoscope.
  Arms: C-MAC group

SUMMARY:
Obesity is associated with difficult intubation rate of 30%, and this study was performed to compare the use of McCoy laryngoscope and C-MAC D-blade video laryngoscope for intubation in obese patients. A total 104 patients with body mass index (BMI) ≥ 35kg/m² scheduled for general anesthesia were randomly assigned to be intubated with McCoy laryngoscope or C-MAC D-blade video laryngoscope. The primary outcome was intubation time, and secondary outcomes were mask ventilation scale, intubation difficulty scale (IDS), percentage of glottis opening (POGO) score, and hemodynamic variables including mean arterial pressure, heart rate and saturation.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status of I-II patients with BMI ≥ 35 kg/m² scheduled for general anesthesia

Exclusion Criteria:

* patients with tracheal diseases, sore throat, neck pain and loose tooth.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Intubation time | The patients were excluded in this study if intubation time was over 90 seconds.
  Timing measurement began when the laryngoscope blade was inserted in patients' mouth and ended when end tidal carbon dioxide tracing was detected in the monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym university sacred heart hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No